CLINICAL TRIAL: NCT03648840
Title: Human Alcohol Seeking Despite Aversion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment paused when our alcohol supplier recalled and suspended manufacture of the product. When production resumed, there was not enough time remaining to successfully resume recruitment. We will examine the outcomes with the existing sample.
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Martin Plawecki, Assistant Professor of Psychiatry, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1709318986; P60AA007611 (NIH)
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: 2 session crossover, random order, single blind
Who Masked: Participant
Masking Description: Subjects are not informed which session will include aversive cues.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher lifetime alcohol drinking (Experimental): Participants with a history of higher lifetime alcohol consumption
  Interventions: Behavioral: Aversive Cue; Behavioral: Neutral Cue
- Lower lifetime alcohol drinking (Experimental): Participants with a lower lifetime alcohol consumption
  Interventions: Behavioral: Aversive Cue; Behavioral: Neutral Cue

INTERVENTIONS:
Behavioral: Aversive Cue — Participants will be exposed to unpleasant pictures and tones during performance of a task to earn alcohol
Behavioral: Neutral Cue — Participants will be exposed to neutral pictures and tones during performance of a task to earn alcohol

SUMMARY:
Prolonged alcohol use results in drinking despite resultant problems and adverse consequences. The investigators propose to test a laboratory model of human seeking despite aversion to use as an early marker of disease onset, and as a tool for study of its neural functional substrates, and identification of effective treatments.

DETAILED DESCRIPTION:
The long-term goal for this project is to establish a model of alcohol seeking despite aversion (SDA) as a platform for the laboratory testing of novel pharmacologic and behavioral interventions that can be used among those with the highest risk, but who have yet to progress to treatment-resistant drinking. The objective of this application is to test SDA across multiple levels of analysis. The investigators consider SDA as an early marker of alcohol use disorder progression that is related to lifetime drinking history, alcohol use disorder risks, and brain physiology. The investigators have completed a pilot study demonstrating that SDA can be objectively quantified via an intravenous alcohol self-administration task, in which operant work for identical incremental alcohol rewards is paired with aversive stimuli. This preliminary data supports the central hypotheses that behavior in the SDA model is attributable to lifetime alcohol exposure, is related to alcohol use disorder risk factors and phenotypes, and reflects alterations in neural system function. In this project, SDA will be measured along with recent and lifetime drinking history, negative affect-based rash action (i.e. negative urgency, including action with respect to alcohol use), and self-rating of the effects of alcohol. The rationale for this work is that it would lead to the first objective, well-validated measure of SDA in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women age 21-55
* Range of lifetime alcohol drinking history from 25 kg to 500 kg, with preference for extremes, plus recent drinking at least 7 drinks/week (women) and 20 drinks/week (men)
* Able to understand and complete questionnaires and procedures in English
* Willing and able to tolerate iv placement
* Right-handed (for fMRI Arm only)

Exclusion Criteria:

* Pregnant or breast-feeding
* Seeking or in treatment for substance use disorder or under court ordered abstinence
* Medications, medical disorders or conditions that could affect study outcome or subject safety
* Positive urine drug screen for amphetamines/methamphetamines, barbiturates, benzodiazepines, cocaine, opiates, or phencyclidine
* Positive breath alcohol (BrAC) reading on arrival at any study visit
* Actively suicidal (within previous year)
* Left-handed or ambidextrous (for fMRI Arm only)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Plawecki, MD, PhD, Principal Investigator — Psychiatry, Indiana University School of Medicine; Melissa A Cyders, PhD, Principal Investigator — Psychology, Indiana University-Purdue University at Indianapolis
Locations (1):
- University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
After publication of the main findings, a de-identified dataset will be made available through direct requests as described above; a statement to this effect will be included in all published manuscripts.
  The current proposal utilizes the Seeking Despite Aversion Task, a newly developed Computer-Assisted Infusion System (CAIS) protocol that integrates delivery of visual stimuli into the Constant Attention Task and optical markers for evoked response potential generation. This task, like other CAIS protocols, will become part of the portfolio of CAIS programs that our lab makes available to other scientists once our specific funded use of this protocol is completed. Modified versions of this protocol could be provided to other investigators prior to completion of this project as long as these projects do not directly compete.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available following final publication of all manuscripts by the component investigators. Earliest date is estimated to be January, 2025.
Access Criteria: Data and Resource Sharing Plan - Indiana Alcohol Research Center (IARC)
  Consistent with its past history, the IARC continues to make available its data and resources to investigators engaged in alcoholism research outside of Indiana University. Detailed procedures are available on request. In brief, investigators must submit a written request specifying in adequate detail the specific resource(s) required and a study protocol indicating the specific aims, scientific rationale, methods and procedure, and analysis of results; a signed IARC Resource Utilization Agreement Form; and for studies involving human subjects, Institutional Review Board (IRB) approval if needed for the proposed study. The request will be reviewed by the IARC Steering Committee. Investigators must agree to acknowledge the Indiana Alcohol Research Center (P60 AA007611) as the source of the resource in all resulting publications.

REFERENCES:
- [Derived] Garrison ACS, Wu W, Cox MR, Haines D, Hays J, Mlungwana MK, Kosobud AEK, Kareken DA, O'Connor S, Plawecki MH, Cyders MA. Aversion-resistant alcohol seeking in the human laboratory. Alcohol Clin Exp Res (Hoboken). 2025 Jul;49(7):1518-1529. doi: 10.1111/acer.70078. Epub 2025 Jul 6. PMID 40618299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general public local to Indianapolis, Indiana. Recruiting methods included flyering, ads run in local publications, and word of mouth. Recruiting period ran from January, 2018 to July, 2022.
Groups:
- Aversive Cue First, Then Neutral Cue; Neutral Cue First, Then Aversive Cue: Participants could earn brief increases in breath alcohol concentration by performing an attention task during two 3-hour IV alcohol infusion sessions scheduled 5-14 days apart. During the Aversive Cue session, participants were exposed to unpleasant pictures and tones during the attention task. During the Neutral Cue session, participants were exposed to neutral pictures and tones during the attention task. Session order was randomly assigned.
Period: First IV Infusion Session
Arm/Group | Aversive Cue First, Then Neutral Cue | Neutral Cue First, Then Aversive Cue
Started | 39 | 48
Completed | 39 | 46
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2
Period: Session 1 to Session 2 Interval
Arm/Group | Aversive Cue First, Then Neutral Cue | Neutral Cue First, Then Aversive Cue
Started | 39 | 46
Completed | 39 | 45
Not Completed | 0 | 1
Not completed — Pandemic | 0 | 1
Period: Second IV Infusion Session
Arm/Group | Aversive Cue First, Then Neutral Cue | Neutral Cue First, Then Aversive Cue
Started | 39 | 45
Completed | 39 | 45
Not Completed | 0 | 0
Period: Session 2 to Imaging Interval
Arm/Group | Aversive Cue First, Then Neutral Cue | Neutral Cue First, Then Aversive Cue
Started | 39 | 45
Completed | 28 | 29
Not Completed | 11 | 16
Not completed — Participant declined fMRI at enrollment | 8 | 11
Not completed — MRI exclusion (left handed) | 3 | 5
Period: fMRI Session
Arm/Group | Aversive Cue First, Then Neutral Cue | Neutral Cue First, Then Aversive Cue
Started | 28 (Planned enrollment for the imaging session was lower than planned enrollment for infusions. Some participants were enrolled in to participate in the infusions who were ineligible for fMRI or who opted out of the fMRI.) | 29 (Planned enrollment for the imaging session was lower than planned enrollment for infusions. Some participants were enrolled in to participate in the infusions who were ineligible for fMRI or who opted out of the fMRI.)
Completed | 28 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The planned primary outcome, reported below, is a comparison between participants with higher versus lower lifetime alcohol drinking. Therefore, baseline characteristics are provided for participants within these two groups.
Groups:
- Higher Lifetime Alcohol Drinking: Participants with a history of higher lifetime alcohol consumption will complete 2 IV alcohol infusion sessions that include aversive or neutral cues.
- Lower Lifetime Alcohol Drinking: Participants with a history of lower lifetime alcohol consumption will complete 2 IV alcohol infusion sessions that include aversive or neutral cues.
- Total: Total of all reporting groups
Arm/Group | Higher Lifetime Alcohol Drinking | Lower Lifetime Alcohol Drinking | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.3 (10.8) | 30.6 (10.5) | 31.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 16 | 23 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 37 | 40 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 24 | 28 | 52
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 40 | 44 | 84

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Exposure to Aversive Cues on IV Alcohol Self-administration
Description: Participants earn 2.5 min exposures to an increase in iv infusion rate (causing a prescribed increase in breath alcohol concentration (BRAC)) by completing repetitions of a constant attention button-pressing task (CAT). The task is designed so that the number of correct CAT trials required increases progressively from 1 (for the first drink) to 380 (for the 20th drink) on an accelerating scale. The dependent measure Breakpoint is defined as the cumulative number of correct and incorrect CAT trials completed when the last drink is earned; in the time allowed possible values ranged from 1 to 800. Effect of the Aversive cue was assessed by calculating a difference score (Breakpoint Aversive Cue-Breakpoint Neutral Cue); the range of possible difference scores was -800 to +800. A positive difference score indicates a higher breakpoint (more alcohol earned) in the Aversive Cue session; a negative number indicates a lower breakpoint (less alcohol earned).
Time Frame: In two infusion sessions, to occur 5-14 days apart
Population: Between subjects design
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Higher Lifetime Alcohol Drinking; Lower Lifetime Alcohol Drinking: Lifetime drinking history is estimated using lifetime drinks per drinking day using a time-line follow back method. Higher and lower drinking groups are defined using the NIH-NIAAA standard: For the Higher drinking group, average lifetime drinks per drinking day was >= 4 for women and 5 for men; for the lower drinking group, average lifetime drinks per drinking day was <4 for women and <5 for men
Arm/Group | Higher Lifetime Alcohol Drinking | Lower Lifetime Alcohol Drinking
Number analyzed (Participants) | 41 | 43
Units on a scale | -6.0 (8.6) | 7.3 (6.9)
Statistical Analysis 1: Comparison: Higher Lifetime Alcohol Drinking vs Lower Lifetime Alcohol Drinking; 2-tailed, unpaired T-test; Test type: Other; p < 0.2, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From enrollment to end of the final study day, usually about 8 weeks.
Groups:
- Aversive Cue: Participants who completed part or all of the Aversive Cue session
- Neutral Cue: Participants who completed part or all of the Neutral Cue session
- fMRI: Participants who completed part or all of the fMRI session
Arm/Group | Aversive Cue | Neutral Cue | fMRI
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/87 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/87 | 0/57
Other Adverse Events (participants affected / at risk) | 3/84 | 4/87 | 3/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aversive Cue (N=84) | Neutral Cue (N=87) | fMRI (N=57)
IV pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) — IV pain during infusions is an anticipated risk
Nausea (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) — Nausea is an anticipated risk of iv infusion of alcohol solutions
Upset by aversive images (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — One subject was upset by the aversive images shown, but chose to continue the session after a short break
Claustrophobia (General disorders) | 0 (0) | 0 (0) | 1 (1) — Claustrophobia in the scanner is an anticipated risk
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) — General discomfort in scanner is an anticipated risk
Nerve Stimulation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Nerve stimulation during imaging is an anticipated risk

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03648840/Prot_SAP_001.pdf
  • Informed Consent Form (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT03648840/ICF_000.pdf